CLINICAL TRIAL: NCT05155670
Title: Hand Motor Rehabilitation Using a Wearable Robotic Device (WRL HX MCP): a Pilot Study
Brief Title: Hand Motor Rehabilitation Using a Wearable Robotic Device (WRL HX MCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Habilis 2020
Record Dates: First submitted 2021-11-21; First posted 2021-12-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hand Injuries
Keywords: Humans; Adult; Diseases, musculoskeletal; Metacarpophalangeal Joints; Range of Motion, Articular; Feasibility Studies; Rehabilitation Research; Robotics; Exoskeleton Device; Wearable Electronic Devices
MeSH Terms: conditions — Hand Injuries; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic therapy (Experimental): All participants will receive a program of robot-assisted rehabilitation exercises., including passive, active-assisive and active MCP Range-of-Motion Exercises, and active bidigital pinching movements in the transparent mode.
  Interventions: Device: WRL HX MCP

INTERVENTIONS:
Device: WRL HX MCP — WRL HX MCP is a non CE marked class IIa medical device designed for clinical application in hand rehabilitation; it consists in a cable-driven robotic MCP orthosis providing flexion-extension of the metacarpo-phalangeal joint. WRL HX MCP features and a series-elastic actuators (SEA) architecture for compliant actuation of MCP flexion-extension and a self-aligning mechanism to absorb human/robot joint axes misplacement. Exoskeleton module is mounted on a dorsal hand support and connected to its electronic box through wires.

SUMMARY:
The purpose of this pilot study is to assess the safety and usability of the WRL HX MCP medical device, a prototypal robotic system for metacarpophalangeal joint mobilization. WRL HX MCP was developed by the Wearable Robotics Laboratory of Scuola Superiore Sant'Anna in a project funded by and in collaboration with INAIL, to fulfil the needs of patients with post-traumatic hand stiffness.

DETAILED DESCRIPTION:
This study aims to:

1. Test the safety and reliability of the WRL HX MCP device for assisting flexion and extension movement of the stiff metacarpophalangeal joint
2. Conduct a preliminary examination of the efficacy of the device in the treatment of joint stiffness to design a subsequent RCT
3. Evaluate the performance of the device in estimating the biomechanical parameters useful for the objective treatment outcome assessment.

Ten injured workers with post-traumatic and/or post-operative index finger MCP stiffness will be enrolled in a clinical trial consisting of one to four sessions of robotic therapy with WRL HX MCP at the INAIL Rehabilitation Center in Volterra.

Pilot testing of the experimental device will include the preliminary goniometric measure of passive and active MCP range of motion (ROM), the selection of the appropriate size of exoskeleton segments to fit user's anthropometry, the robotic assessment of ROM, force and torque trajectories of MCP joint, a program of robot-assisted passive and active MCF mobilization and a final clinical and robotic reassessment of joint ROM. The session will last about 1 hour and all exercises will be administered by a trained physical therapist supported by two members of the engineering team; pain level will be assessed at baseline and after each mobilization sequence; patient feedback will be recorded about the usability of the device in term of comfort, wearability, user safety, and overall satisfaction.

For Aim 1, the Safety and Reliability of the device will be evaluated in terms of the number of adverse events and malfunctions occurring during the study session.

For Aim 2, the efficacy of robot-assisted mobilization modes will be assessed by means of the longitudinal analysis of pre- and post-treatment measurements of MCP range of motion and pain intensity level, the flexion peak torque evaluation and the final administration of an ad-hoc satisfaction questionnaire.

For aim 3, the performance of WRL HX MCP will be studied by comparing the robotic MCP angle estimation with the measurements from a motion capture system.

ELIGIBILITY:
Inclusion Criteria:

* history of traumatic hand injury or post-traumatic hand surgery
* hand size allowing to achieve proper exoskeleton fit
* NRS pain score in the 1-5 range

Exclusion Criteria:

* cognitive or linguistic ability insufficient to understand instructions
* cardiac implanted electronic devices
* open skin at the level of the patient-device interface
* absence of contraindications for finger joints mobilisation
* current or prior history of malignancy
* pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Feasibility indicator: completion of study procedures | through study completion, an average of 1 year
  Percent of participants for whom study procedures were completed successfully
Feasibility indicator: patient acceptability | After the robotic therapy session; the total expected time for the session is about 90 minutes.
  Clinician-generated questionnaire to investigate patients' impressions about the physical interaction with the robotic device
Feasibility indicator: reliability evaluated through the number of device malfunctions | through study completion, an average of 1 year
  The physiotherapist is required to report any malfunctions occurring during the study in regard to the use of WRL HX MCP

SECONDARY OUTCOMES:
Goniometric measure of MCP Active Range of Motion (AROM) | at baseline and immediately after the robotic therapy session.
  The physiotherapist measures the MCP joint angles in maximum active flexion and extension using a short-arm goniometer
Goniometric measure of MCP Passive Range of Motion (PROM) | at baseline and immediately after the robotic therapy session
  The physiotherapist measures the MCP joint angles in maximum passive flexion and extension using a short-arm goniometer
Robotic measure of MCP Active Range of Motion (AROM) | at baseline and immediately after the robotic therapy session
  MCP joint maximum active flexion and extension range of motion is registered while the device and human joint are coupled together, using WRL HX MCP set in a transparent mode as an evaluation tool, without any manual assistance.
Robotic measure of MCP passive Range of Motion (PROM) | at baseline and immediately after the robotic therapy session
  MCP joint maximum passive flexion and extension range of motion is registered while the device and human joint are coupled together, using WRL HX MCP set in a transparent mode as an evaluation tool, with manual assistance from the therapist.
Robotic estimation of MCP joint flexion peak torque | during robot-in-charge mobilization sequences
  MCP joint flexion peak torque is evaluated by the exoskeleton torque joint sensor during the robot-in-charge mobilization sequences
Numeric Pain Rating Scale (NPRS) | at baseline and after each of the two series of joint mobilization exercises, lasting up to 30 minutes each.
  NPRS is an 11-point scale for patient self-reporting of pain, with 0 being "no pain" and 10 being "the worst pain imaginable"
Safety evaluated through the number of adverse events | through study completion, an average of 1 year
  The physiotherapist is required to report any adverse events occurring during the study in regard to the use of WRL HX MCP

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Taglione, MD, Principal Investigator — INAIL - Centro di Riabilitazione Motoria di Volterra; Simona Crea, PhD, Study Director — The BioRobotics Institute, Scuola Superiore Sant'Anna
Locations (1):
- INAIL - Centro di Riabilitazione Motoria di Volterra, Volterra, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kollitz KM, Hammert WC, Vedder NB, Huang JI. Metacarpal fractures: treatment and complications. Hand (N Y). 2014 Mar;9(1):16-23. doi: 10.1007/s11552-013-9562-1. PMID 24570632
- [Background] Evans RB. Managing the injured tendon: current concepts. J Hand Ther. 2012 Apr-Jun;25(2):173-89; quiz 190. doi: 10.1016/j.jht.2011.10.004. Epub 2012 Feb 11. PMID 22326362
- [Background] Ye L, Kalichman L, Spittle A, Dobson F, Bennell K. Effects of rehabilitative interventions on pain, function and physical impairments in people with hand osteoarthritis: a systematic review. Arthritis Res Ther. 2011 Feb 18;13(1):R28. doi: 10.1186/ar3254. PMID 21332991
- [Background] Metcalf C, Adams J, Burridge J, Yule V, Chappell P. A review of clinical upper limb assessments within the framework of the WHO ICF. Musculoskeletal Care. 2007 Sep;5(3):160-73. doi: 10.1002/msc.108. PMID 17610309
- [Background] Krebs HI, Volpe BT. Rehabilitation robotics. Handb Clin Neurol. 2013;110:283-94. doi: 10.1016/B978-0-444-52901-5.00023-X. PMID 23312648
- [Background] M. Cempini, M. Cortese and N. Vitiello,
- [Background] Soekadar SR, Witkowski M, Gomez C, Opisso E, Medina J, Cortese M, Cempini M, Carrozza MC, Cohen LG, Birbaumer N, Vitiello N. Hybrid EEG/EOG-based brain/neural hand exoskeleton restores fully independent daily living activities after quadriplegia. Sci Robot. 2016 Dec 6;1(1):eaag3296. doi: 10.1126/scirobotics.aag3296. Epub 2016 Nov 16. PMID 33157855
- [Background] Marconi, D., Baldoni, A., McKinney, Z., Cempini, M., Crea, S., & Vitiello, N. (2019). A novel hand exoskeleton with series elastic actuation for modulated torque transfer. Mechatronics, 61, 69-82. https://doi.org/10.1016/j.mechatronics.2019.06.001
- [Background] Carpinella I, Mazzoleni P, Rabuffetti M, Thorsen R, Ferrarin M. Experimental protocol for the kinematic analysis of the hand: definition and repeatability. Gait Posture. 2006 Jun;23(4):445-54. doi: 10.1016/j.gaitpost.2005.05.001. Epub 2005 Jun 22. PMID 15978812
- [Background] A. Chiri et al.,
- [Background] Cempini M, Marzegan A, Rabuffetti M, Cortese M, Vitiello N, Ferrarin M. Analysis of relative displacement between the HX wearable robotic exoskeleton and the user's hand. J Neuroeng Rehabil. 2014 Oct 18;11:147. doi: 10.1186/1743-0003-11-147. PMID 25326697
- [Derived] Peperoni E, Trigili E, Capotorti E, Capitani SL, Fiumalbi T, Pettinelli F, Grandi S, Rapalli A, Lentini G, Creatini I, Vitiello N, Taglione E, Crea S. Post-traumatic hand rehabilitation using a powered metacarpal-phalangeal exoskeleton: a pilot study. J Neuroeng Rehabil. 2024 Dec 19;21(1):214. doi: 10.1186/s12984-024-01511-w. PMID 39702346